CLINICAL TRIAL: NCT03840993
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Assess the Safety and Efficacy of MT-2990 in Women With Endometriosis Experiencing Endometrial Related Pain
Brief Title: Safety and Efficacy Study of MT-2990 in Women With Endometriosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT-2990-A01
Record Dates: First submitted 2019-02-04; First posted 2019-02-15 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Related Pain
Keywords: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MT-2990 (Experimental): MT-2990, over 16 weeks
  Interventions: Drug: MT-2990
- Placebo (Placebo Comparator): Placebo, over 16 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT-2990 — over 16 weeks
  Arms: MT-2990
Drug: Placebo — over 16 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of MT-2990 for treatment of moderate to severe endometriosis-related pain in women with surgically diagnosed endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent to participate in this study
* Agree to approximately 30-90 day washout interval of hormonal therapies, if applicable
* Have a history of regular menstrual cycles
* Have a body mass index < 45 kg/m^2 (inclusive)
* Have documented surgical/laparoscopy diagnosis of endometriosis with 10 years
* Agree to use 2 forms of nonhormonal contraception throughout the study
* In the Investigator's opinion, subject is able to understand the nature of the study and any risk involved in participation, and is willing to cooperate and comply with the protocol restrictions and requirements including transvaginal ultrasound.
* Have moderate to severe endometrial related pain

Exclusion Criteria:

* Subject is pregnant, breast feeding, or planning a pregnancy.
* Subject is < 6 months postpartum, postabortion, or post-pregnancy.
* Willing to remove a hormonal intrauterine device (IUD) at least 30 days prior to screening. (Non hormonal IUDs do not have to be removed)
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT) , or total bilirubin ≥ 2.0 × upper limit of normal (ULN) above the reference range
* Have immunosuppression due to underlying medical condition
* Corrected QT interval using Fridericia's formula (QTcF) or Corrected QT interval using Bazett's formula (QTcB) ≥ 450 msec or clinically important abnormal findings on the ECG
* Subject is not up-to-date on breast screening according to current guidelines.
* Has a surgical history of hysterectomy, bilateral oophorectomy and any other recent major surgery
* Subject is required more than 2 weeks of continuous use of prohibited long-acting narcotic or immediate release narcotic for treatment of endometriosis-associated pain.
* Have chronic pelvic pain for nonendometriosis related causes, which require systemic pharmaceutical chronic therapy for pain
* Have other chronic pain syndrome which require chronic analgesic or other chronic therapy
* Have a clinically significant gynecologic condition identified on the transvaginal ultrasound (TVU) (e.g., complex ovarian cyst > 3 cm or simple ovarian cyst > 5 cm, clinically significant endometrial pathology, single fibroid ≥ 4 cm or multiple (> 4) fibroids that measure ≥ 2 cm or symptomatic submucosal fibroid of any size
* Have a current history of undiagnosed abnormal genital bleeding

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2021-05-13 (Actual); Study Completion 2021-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Head of Medical Science, Study Director — Tanabe Pharma America, Inc.
Locations (51):
- United States (51):
  - Precision Trials, Phoenix, Arizona
  - Northern California Research Corporation, Sacramento, California
  - Ageless and Beautiful Medical Spa, San Diego, California
  - Precision Research Institute, San Diego, California
  - The Lundquist Institute at Harbor-UCLA Medical Center, Torrance, California
  - Clinical Physiology Associates - Fort Myers, Fort Myers, Florida
  - AGA Clinical Trials, Hialeah, Florida
  - Kendall South Medical Center, Hialeah, Florida
  - South Florida Clinical Trials, Hialeah, Florida
  - Altus Research, Lake Worth, Florida
  - Axcess Medical Research, Loxahatchee Groves, Florida
  - Health and Life Research Institute, Miami, Florida
  - Ivetmar Medical Group, Miami, Florida
  - Future Care Solution, Miami, Florida
  - Advanced Medical Research Institute, Miami, Florida
  - South Florida Research Phase I-IV, Miami Springs, Florida
  - American Research Centers of Florida, Pembroke Pines, Florida
  - Agile Clinical Research Trials, Alpharetta, Georgia
  - Medi-Sense, Atlanta, Georgia
  - NuDirections Clinical Research, Dunwoody, Georgia
  - Drug Studies America - Marietta, Marietta, Georgia
  - Clinical Research Prime, Idaho Falls, Idaho
  - Rosemark Women Care Specialists, Idaho Falls, Idaho
  - Advanced Clinical Research - Idaho, Meridian, Idaho
  - The Advanced Gynecologic Surgery Institute, Park Ridge, Illinois
  - GTC Research, Shawnee Mission, Kansas
  - Clinical Trials Management - Covington Northshore Office, Covington, Louisiana
  - Southern Clinical Research Associates, Metairie, Louisiana
  - Omni Fertility and Laser Institute, Shreveport, Louisiana
  - Continental Clinical Solutions, Towson, Maryland
  - Saginaw Valley Medical Research Group/Women's OB-GYN, Saginaw, Michigan
  - Albuquerque Clinical Trials, Albuquerque, New Mexico
  - Manhattan Medical Research, New York, New York
  - Carolina Women's Research and Wellness Clinic, Durham, North Carolina
  - Unified Women's Clinical Research - Raleigh, Raleigh, North Carolina
  - PMG Research of Rocky Mount, Rocky Mount, North Carolina
  - Lyndhurst Gynecologic Associates, Winston-Salem, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Aventive Research - Colombus, Columbus, Ohio
  - North Star Medical Research, Middleburg Heights, Ohio
  - ClinEdge - Fusion Clinical Research of Spartanburg, Spartanburg, South Carolina
  - Wake Research Associates, Chattanooga, Tennessee
  - Precision Research Institute - Houston, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Biopharma Informatic - Houston, Houston, Texas
  - Discovery Clinical Trials, San Antonio, Texas
  - Physician's Research Options (PRO), Draper, Utah
  - Physician's Research Options (PRO), Pleasant Grove, Utah
  - Wasatch Clinical Research, Salt Lake City, Utah
  - Health Research of Hampton Roads, Newport News, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | MT-2990
Started | 39 | 37
Completed | 30 | 30
Not Completed | 9 | 7
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 4 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Pregnancy | 0 | 1
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Neutrophil count decrease, COVID-19 | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MT-2990 | Total
Number analyzed (Participants) | 39 | 37 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.9 (8.3) | 32.7 (7.6) | 33.8 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 37 | 76
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20 | 15 | 35
  Not Hispanic or Latino | 19 | 22 | 41
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline to Week 16 in Nonmenstrual Pelvic Pain Using a Pain Scale Ranges From 0 (None) to 3 (Severe)
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 32 | 29
units on a scale | -0.28 (0.12) | -0.63 (0.12)

2. Secondary Outcome: Mean Change From Baseline to Week 16 in Dysmenorrhea Using a Pain Scale Ranges From 0 (None) to 3 (Severe)
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 32 | 29
units on a scale | -0.47 (0.15) | -0.68 (0.16)

3. Secondary Outcome: Mean Change From Baseline to Week 16 in Dyspareunia Using a Pain Scale Ranges From 0 (None) to 3 (Severe)
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 22 | 24
units on a scale | -0.38 (0.19) | -0.57 (0.18)

4. Secondary Outcome: Mean Change From Baseline to Week 16 in Non-Menstrual Pelvic Pain (NMPP) Using a Pain Scale Ranges From 0 (no Pain) to 10 (Worst Pain)
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 32 | 29
units on a scale | -1.05 (0.37) | -2.33 (0.39)

5. Secondary Outcome: Mean Change From Baseline to Week 16 in Dysmenorrhea Using a Pain Scale Ranges From 0 (no Pain) to 10 (Worst Pain)
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 32 | 29
units on a scale | -1.33 (0.48) | -2.28 (0.5)

6. Secondary Outcome: Mean Change From Baseline to Week 16 in Dyspareunia Using a Pain Scale Ranging From 0 (no Pain) to 10 (Worst Pain)
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 19 | 21
units on a scale | -1.32 (0.56) | -2.74 (0.52)

7. Secondary Outcome: Mean Change From Baseline Through Week 16 in the Number of Any Analgesic Pills Used
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Least Squares Mean (Standard Error); unit: pills
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 28 | 27
pills | -0.33 (0.09) | -0.27 (0.09)

8. Secondary Outcome: Mean Change From Baseline Through Week 16 in the Number of Opioid Pills Used
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Least Squares Mean (Standard Error); unit: Pills
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 29 | 27
Pills | -0.01 (0.02) | -0.04 (0.02)

9. Secondary Outcome: Time to Use of Rescue Medication (Analgesic)
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 7 | 7
days | 42.0 [42.0 to 42.0] | 19.0 [19.0 to 19.0]

10. Secondary Outcome: Percentage of NMPP Responders From Baseline Through Week 16 Using a Pain Scale That Ranges From 0 (None) to 3 (Severe)
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Number; unit: percentage of NMPP responders
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 32 | 29
percentage of NMPP responders | 34.4 | 55.2

11. Secondary Outcome: Percentage of Dysmenorrhea Responders From Baseline Through Week 16 Using a Pain Scale That Ranges From 0 (None) to 3 (Severe)
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Number; unit: percentage of dysmenorrhea responders
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 32 | 29
percentage of dysmenorrhea responders | 34.4 | 37.9

12. Secondary Outcome: Percentage of Dyspareunia Responders From Baseline Through Week 16 Using a Pain Scale That Ranges From None (0) to 3 (Severe)
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Number; unit: percentage of dyspareunia responders
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 22 | 24
percentage of dyspareunia responders | 36.4 | 37.5

13. Secondary Outcome: Mean Percentage Change From Baseline Through Week 16 in Nonmenstrual Pelvic Pain Using a Pain Scale That Ranges From 0 (None) to 3 (Severe)
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Least Squares Mean (Standard Error); unit: mean percentage change
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 32 | 29
mean percentage change | -18.87 (7.48) | -37.29 (7.86)

14. Secondary Outcome: Mean Percentage Change From Baseline Through Week 16 in Dysmenorrhea Using a Pain Scale That Ranges From 0 (None) to 3 (Severe)
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Least Squares Mean (Standard Error); unit: Mean percentage change
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 31 | 29
Mean percentage change | -21.92 (7.54) | -30.95 (7.76)

15. Secondary Outcome: Mean Percentage Change From Baseline Through Week 16 in Dyspareunia Using a Pain Scale That Ranges From 0 (None) to 3 (Severe)
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Least Squares Mean (Standard Error); unit: Mean percentage change
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 22 | 24
Mean percentage change | -26.95 (13.18) | -20.88 (12.48)

16. Secondary Outcome: Percentage of NMPP Responders From Baseline Through Week 16 Using a Pain Scale That Ranges From 0 (no Pain) to 10 (Worst Pain Ever)
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Number; unit: percentage of NMPP responders
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 32 | 29
percentage of NMPP responders | 25.0 | 48.3

17. Secondary Outcome: Percentage of Dysmenorrhea Responders From Baseline Through Week 16 Using a Pain Scale That Ranges From 0 (no Pain) to 10 (Worst Pain Ever)
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Number; unit: percentage of dysmenorrhea responders
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 32 | 29
percentage of dysmenorrhea responders | 34.4 | 51.7

18. Secondary Outcome: Percentage of Dyspareunia Responders From Baseline Through Week 16 Using a Pain Scale That Ranges From 0 (no Pain) to 10 (Worst Pain Ever)
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Number; unit: percentage of dyspareunia responders
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 19 | 21
percentage of dyspareunia responders | 31.6 | 47.6

19. Secondary Outcome: Mean Percentage Change From Baseline Through Week 16 in Nonmenstrual Pelvic Pain Using a Pain Scale That Ranges From 0 (no Pain) to 10 (Worst Pain Ever)
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Least Squares Mean (Standard Error); unit: Mean percentage change
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 39 | 36
Mean percentage change | -21.2 (6.72) | -43.07 (7.05)

20. Secondary Outcome: Mean Percentage Change From Baseline Through Week 16 in Dysmenorrhea Using a Pain Scale That Ranges From 0 (no Pain) to 10 (Worst Pain Ever)
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Least Squares Mean (Standard Error); unit: Mean percentage change
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 32 | 29
Mean percentage change | -18.54 (7.12) | -31.37 (7.48)

21. Secondary Outcome: Mean Percentage Change From Baseline Through Week 16 in Dyspareunia Using a Pain Scale That Ranges From 0 (no Pain) to 10 (Worst Pain Ever)
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Least Squares Mean (Standard Error); unit: Mean percentage change
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 19 | 21
Mean percentage change | -29.04 (10.18) | -40.8 (9.4)

22. Secondary Outcome: Number of Responders Using Global 7-point Scale
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 30 | 31
Participants | 12 | 18

23. Secondary Outcome: Percentage of Responders Using Global 7-point Scale
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Number; unit: Percentage of responders
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 30 | 31
Percentage of responders | 40.0 | 58.1

24. Secondary Outcome: Mean Change From Baseline to Weeks 4, 8, 12 and 16 on the Pain Dimension of a Scale Ranging From 100 (Worst) to 0 (Best)
Time Frame: From Baseline to Weeks 4, 8, 12, and 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 39 | 36
units on a scale
  Change from Baseline at Week 4 | -15.58 (3.27) | -19.32 (3.51)
  Change from Baseline at Week 8 | -19.48 (3.56) | -28.60 (3.76)
  Change from Baseline at Week 12 | -20.03 (3.89) | -34.12 (3.99)
  Change from Baseline at Week 16 | -22.55 (3.66) | -33.55 (3.78)

25. Secondary Outcome: Number of Responders Using Endometriosis Specific 7-point Scale
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 30 | 31
Participants | 14 | 19

26. Secondary Outcome: Percentage of Responders Using Endometriosis Specific 7-point Scale
Time Frame: Baseline to Week 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Number; unit: percentage of responders
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 30 | 31
percentage of responders | 46.7 | 61.3

27. Secondary Outcome: Mean Change From Baseline to Weeks 4, 8, 12, and 16 on the Control and Powerlessness Dimension of a Scale Ranging From 100 (Worst) to 0 (Best)
Time Frame: From Baseline to Weeks 4, 8, 12, and 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 37 | 35
units on a scale
  Change from Baseline at Week 4 | -19.80 (3.68) | -24.39 (4.03)
  Change from Baseline at Week 8 | -25.47 (4.42) | -33.78 (4.67)
  Change from Baseline at Week 12 | -26.66 (5.24) | -38.03 (5.42)
  Change from Baseline at Week 16 | -25.27 (5.02) | -35.80 (5.23)

28. Secondary Outcome: Mean Change From Baseline to Weeks 4, 8, 12, and 16 on the Emotional Well-Being Dimension of a Scale Ranging From 100 (Worst) to 0 (Best)
Time Frame: From Baseline to Weeks 4, 8, 12, and 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 37 | 35
units on a scale
  Change from Baseline at Week 4 | -13.31 (3.03) | -13.06 (3.25)
  Change from Baseline at Week 8 | -16.54 (3.26) | -19.01 (3.42)
  Change from Baseline at Week 12 | -15.50 (3.54) | -23.52 (3.57)
  Change from Baseline at Week 16 | -18.17 (3.37) | -23.75 (3.47)

29. Secondary Outcome: Mean Change From Baseline to Weeks 4, 8, 12, and 16 on the Social Support Dimension of a Scale Ranging From 100 (Worst) to 0 (Best)
Time Frame: From Baseline to Weeks 4, 8, 12, and 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 37 | 35
units on a scale
  Change from Baseline at Week 4 | -13.77 (3.66) | -12.21 (3.94)
  Change from Baseline at Week 8 | -22.28 (4.00) | -17.85 (4.21)
  Change from Baseline at Week 12 | -21.35 (4.74) | -23.45 (4.83)
  Change from Baseline at Week 16 | -19.28 (4.50) | -24.52 (4.66)

30. Secondary Outcome: Mean Change From Baseline to Weeks 4, 8, 12, and 16 on the Self-Image Dimension of a Scale Ranging From 100 (Worst) to 0 (Best)
Time Frame: From Baseline to Weeks 4, 8, 12, and 16
Population: Overall Number of Participants Analyzed is all participants with data available in Intent To Treat (ITT) population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | MT-2990
Number analyzed (Participants) | 37 | 35
units on a scale
  Change from Baseline at Week 4 | -17.39 (3.90) | -14.65 (4.20)
  Change from Baseline at Week 8 | -23.20 (4.02) | -21.01 (4.23)
  Change from Baseline at Week 12 | -17.65 (4.59) | -26.45 (4.54)
  Change from Baseline at Week 16 | -19.42 (4.53) | -27.55 (4.65)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Day 1 through to the end of the 16-week double-blind treatment phase.
Arm/Group | Placebo | MT-2990
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/39 | 1/37
Other Adverse Events (participants affected / at risk) | 22/39 | 23/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=39) | MT-2990 (N=37)
Abortion induced (Surgical and medical procedures) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=39) | MT-2990 (N=37)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 4 | 1
Toothache (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Axillary pain (General disorders) | 0 | 1
Catheter site swelling (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Fatigue (General disorders) | 3 | 2
Infusion site pain (General disorders) | 0 | 2
Injection site haemorrhage (General disorders) | 0 | 1
Pain (General disorders) | 0 | 2
Pyrexia (General disorders) | 0 | 1
Bacterial vaginosis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 1
Corona virus infection (Infections and infestations) | 0 | 2
Cystitis (Infections and infestations) | 2 | 0
Localised infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1
Urinary tract infection (Infections and infestations) | 2 | 4
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood cholesterol increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 3
Blood triglycerides increased (Investigations) | 1 | 0
Coronavirus test positive (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Urine analysis abnormal (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Ageusia (Nervous system disorders) | 0 | 2
Anosmia (Nervous system disorders) | 0 | 2
Clonic convulsion (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 2
Meralgia paraesthetica (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Mood swings (Psychiatric disorders) | 0 | 1
Nightmare (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Urge incontinence (Renal and urinary disorders) | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0
Breast cyst (Reproductive system and breast disorders) | 0 | 1
Breast tenderness (Reproductive system and breast disorders) | 1 | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 | 1
Hydrosalpinx (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0
Nipple pain (Reproductive system and breast disorders) | 0 | 1
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0
Flushing (Vascular disorders) | 0 | 1
Hot flush (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2020-03-04): https://cdn.clinicaltrials.gov/large-docs/93/NCT03840993/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/93/NCT03840993/SAP_001.pdf